CLINICAL TRIAL: NCT05089045
Title: A Clinical Study to Evaluate the Immunogenicity and Safety of Recombinant New Coronavirus Vaccine (CHO Cells) After Vaccination With Two Inactivated Vaccine in Healthy People Aged 18 and Above
Brief Title: Immunogenicity and Safety Evaluation of Recombinant Novel Coronavirus Vaccine (CHO Cells) in Enhancing Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LKM-2021-NCV04
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Coronavirus Disease 2019
Keywords: Recombinant Novel Coronavirus Vaccine
MeSH Terms: conditions — COVID-19 | interventions — Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Population Ⅰ (Experimental)
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group

INTERVENTIONS:
Biological: Recombinant new coronavirus vaccine (CHO cell) group — Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).

SUMMARY:
Popular topic: Clinical study on immunogenicity and safety evaluation of sequentially enhanced immunity with recombinant Novel Coronavirus vaccine (CHO cells) Research purpose:Main purpose:To evaluate the immunogenicity of recombinant Novel Coronavirus vaccine (CHO cells) after sequential booster immunization in populations vaccinated with two doses of marketed Novel Coronavirus inactivated vaccine.Secondary purpose:To evaluate the safety of recombinant Novel Coronavirus vaccine (CHO cells) after sequential booster immunization in populations vaccinated with two doses of marketed Novel Coronavirus inactivated vaccine.

Overall design:An open experimental design was used in this study Study population:The study involved people 18 years of age and older. Test groups: All subjects recruited must have received two doses of Novel Coronavirus inactivated vaccine for 3 to 13 months (the interval between booster and basic immunization is divided into 3 groups:120 subjects at 3-4 months (91-120 days), 6-8 months (181-240 days) and 11-13 months (331-390 days) were vaccinated with one dose of recombinant Novel Coronavirus vaccine (CHO cells).

DETAILED DESCRIPTION:
Overall design: An open experimental design was adopted in this study, and 360 subjects were planned to be enrolled.To evaluate the immunogenicity and safety of recombinant Novel Coronavirus vaccine (CHO cells) after sequential booster immunization in populations vaccinated with two doses of marketed Novel Coronavirus inactivated vaccine.

Intervention: This study involved people 18 years of age and older.All subjects recruited must have received two doses of Novel Coronavirus inactivated vaccine for 3 to 13 months (the interval between booster and basic immunization is divided into 3 groups:120 subjects at 3-4 months (91-120 days), 6-8 months (181-240 days) and 11-13 months (331-390 days) were vaccinated with one dose of recombinant Novel Coronavirus vaccine (CHO cells).

Immunogenicity observation:

Blood samples were collected from all subjects before and 14 days after experimental vaccine vaccination for humoral immunoassay.

Safety observation:

AE and SAE:

Collect all adverse events (AE) at least 30 minutes after vaccination, all AE (both solicitation and non-solicitation AE) from 0 to 7 days, and all AE (non-solicitation AE) from 8 to 30 days;All serious adverse events (SAE) within 1 month after vaccination with the experimental vaccine were collected.

1. Solicitation AE (the following events occurring within 0-7 days after vaccination with experimental vaccine) :Adverse events at the inoculation site (local) : pain, itching, redness, swelling, rash, induration; Non-inoculated site (systemic) adverse events: fever, headache, fatigue/fatigue, diarrhea, nausea, vomiting, muscle pain (non-inoculated site), acute allergic reaction, cough.
2. Vital signs and physical examination:All subjects were assessed for vital signs (blood pressure, axillary body temperature, pulse) during screening and axillary body temperature before trial vaccination.

   All subjects underwent physical examination (skin, cardiopulmonary auscultation) during the screening period.
3. Collection of pregnancy events:Women of childbearing age should undergo a urine pregnancy test before enrollment (on the day of vaccination).

   Pregnancy events occurring within 1 month after trial vaccination were collected.
4. ADE/VED (Antibody enhancement/vaccine Enhancement) Risk Monitoring:After receiving the experimental vaccine, if the subject is diagnosed with COVID-19, he/she should go to the hospital for hospitalization or be isolated in accordance with the local epidemic prevention and control requirements.A special investigation will be conducted for severe/critical/fatal cases, and the existence of ADE/VED will be analyzed based on the results of the special investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 and over with full civil capacity who can provide vaccination information proving that they have received two doses of Novel Coronavirus inactivated vaccine (Vero cells) in the last 3-13 months;
2. Subjects voluntarily participate in the study, sign informed consent, provide valid identification, understand and comply with the requirements of the study protocol;
3. Fertile men and women of reproductive age did not have sex from day 1 of the last menstrual cycle to day 1 of the study, or did not have sex with an effective contraceptive method and did not experience contraceptive failure (examples of contraceptive failure include male condom rupture during sex).Subjects also agreed to use effective contraception from the time of signing informed consent to 1 month after trial vaccination.

Exclusion Criteria:

1. History of confirmed or asymptomatic coronavirus infection or positive nucleic acid test of novel Coronavirus infection;
2. SARS virus history;
3. Fever caused by any reason (such as cold, local inflammation, tumor, rheumatic immune disease, etc.) within 72 hours before enrollment, or armpit temperature ≥37.3℃ on the day of enrollment;
4. history of severe allergic to any vaccine, or to test the vaccine's active ingredient, any a kind of active ingredients, use of material in the production process, including aluminum has a history of severe allergic, for example: the acute allergic reaction and allergic shock, allergic laryngeal edema, thrombocytopenic purpura, allergic purpura, difficulty breathing, angioneurotic oedema, etc;
5. Persons suffering from the following diseases:

   ① Patients with stroke and encephalitis in the acute stage, patients with immune-related neurological diseases (such as myomyelitis, Guillanbarre syndrome, demyelinating disease, myasthenia gravis, etc.) that are not controlled, patients with epilepsy and severe mental illness, and patients with other neurological diseases that are not controlled;

   ② Patients with acute respiratory infection, acute attack of chronic obstructive pulmonary disease, acute attack of bronchial asthma or clinical uncontrolled stage, acute stage of pleural disease, etc.;

   ③ systolic blood pressure ≤90mmHg and/or diastolic blood pressure ≤60mmHg of unknown cause;Hypertension treated with lifestyle adjustment and/or medication, systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg;Severe coronary heart disease, arrhythmia, heart rate less than 60 beats/min or more than 100 beats/min;Serious heart valve disease, aortic dissection, venous thrombosis;Patients with severe heart failure;Severe arrhythmia, or patients with acute coronary syndrome, acute aortic syndrome, etc.;

   ④ patients with acute pancreatitis, acute intestinal obstruction, acute hepatitis, patients with gastrointestinal bleeding symptoms, active stage of inflammatory bowel disease, active stage of chronic hepatitis, active stage of tuberculosis, etc.;

   ⑤ Patients with acute urinary and reproductive system infection, patients with severe kidney disease (uncontrolled acute and chronic nephritis, patients who are using glucocorticoids, immunosuppressants or biological agents, patients with acute renal insufficiency or chronic kidney disease stage 3 or more namely glomerular filtration rate eGFR<60ml/min);

   ⑥ Diabetes patients with acute complications (remunerative acidosis, hyperotonic state, lactic acidosis) or with the above acute complications recovered less than 2 weeks;Fasting blood glucose > 13.9 mmol/L;Hypothyroidism TSH & GT;10 µ IU/L, with T3 and T4 lower than normal;Patients with uncontrolled hyperthyroidism or hyperthyroidism;

   ⑦ lymphoproliferative disease uncontrolled period, aplastic anemia not alleviated period, primary immune thrombocytopenia (ITP) activity period, coagulation disease uncontrolled period and other patients;

   ⑧ Was immune system disease (systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, sjogren's syndrome, etc.) in active patients, patients with congenital or acquired immunodeficiency, clear merge opportunistic infections or malignant tumors uncontrolled HIV infection, patients with lymphoma, leukemia or autoimmune inflammatory disease;

   ⑨ Patients with malignant tumor undergoing chemotherapy, radiotherapy, and immunotherapy before and after surgery;Patients with organ transplant status;

   ⑩ Patients with acute stage of severe allergic rhinitis, acute and chronic eczema or urticaria with obvious symptoms and signs, or patients with other skin symptoms;

   ⑪ The absence of spleen or history of splenic surgery;
6. Receive immunomodulators within 6 months, such as immunosuppressive doses of glucocorticoids (dose reference: equivalent to prednisone 20mg/ day, over a week);Or monoclonal antibodies;Or thymosin;Or interferon;However, topical use (such as ointments, eye drops, inhalants or nasal sprays) is allowed;
7. Have received blood or blood-related products, including immunoglobulin (including rabies immunoglobulin and tetanus immunoglobulin), within 3 months prior to experimental vaccine vaccination;Or planned use of the experimental vaccine within 1 month of vaccination;
8. For those who have received rabies vaccine and tetanus vaccine and have not completed the course of vaccination, other subunit vaccines and inactivated vaccines shall be injected within 14 days before the experimental vaccine inoculation, and other live attenuated vaccines shall be injected within 30 days before the experimental vaccine inoculation;
9. Women who are breastfeeding or pregnant (including women of childbearing age who have positive urine pregnancy test) or who plan to have a pregnancy within 1 month of the test vaccine or their partners;
10. Have participated in or are participating in other COVID-19 related clinical trials, in addition to completing two doses of inactivated novel Coronavirus vaccine in the past 3-13 months;
11. The Investigator believes that the subject has any disease or condition that may place the subject at unacceptable risk;Subjects cannot meet the requirements of the program;Conditions that interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
The number of adverse events after intramuscular injection | 1 months after full vaccination
  The main observation methods of adverse reactions mainly include local reactions and systemic reactions at the administration site.
Immunogenic end point | 14 days after vaccination
  GMT and positive rate of SARS-COV-2 neutralizing antibody 14 days after vaccination with recombinant Novel Coronavirus vaccine (CHO cells)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No